CLINICAL TRIAL: NCT03765801
Title: Phase I, Single-center Study to Explore the Relative Bioavailability and the Effect of Food on the Bioavailability of Prolonged Release Tablets Compared to Immediate Release Capsules Each Containing 60 mg of GRTA9906 in 20 Healthy Female Volunteers
Brief Title: A Clinical Study in Healthy Women Which Aims to Explore the Intestinal Uptake of Two Different Tablets of GRTA9906 Into the Body and the Effect of Food on it
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP9906/06
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Pain; Neuropathic Pain; Chronic Pain; Visceral Pain
MeSH Terms: conditions — Pain; Neuralgia; Chronic Pain; Visceral Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GRTA9906 60 mg PR tablet (fed) (Experimental): Participants will receive two 60 mg GRTA9906 PR matrix tablets under fed conditions after consumption of a high-fat and high-calorie test meal.
  Interventions: Drug: GRTA9906 60 mg PR tablet
- GRTA9906 60 mg PR tablet (fasting) (Experimental): Participants will receive two 60 mg GRTA9906 PR matrix tablets under fasting conditions (10 hours before dosing until 4.5 hours after dosing).
  Interventions: Drug: GRTA9906 60 mg PR tablet
- GRTA9906 60 mg IR capsule (fed) (Experimental): Participants will receive two 60 mg GRTA9906 IR capsules under fed conditions after consumption of a high-fat and high-calorie test meal.
  Interventions: Drug: GRTA9906 60 mg IR capsule
- GRTA9906 60 mg IR capsule (fasting) (Experimental): Participants will receive two 60 mg GRTA9906 IR capsules under fasting conditions (10 hours before dosing until 4.5 hours after dosing).
  Interventions: Drug: GRTA9906 60 mg IR capsule

INTERVENTIONS:
Drug: GRTA9906 60 mg PR tablet — GRTA9906 60 mg PR tablet
  Arms: GRTA9906 60 mg PR tablet (fasting); GRTA9906 60 mg PR tablet (fed)
Drug: GRTA9906 60 mg IR capsule — GRTA9906 60 mg IR capsule
  Arms: GRTA9906 60 mg IR capsule (fasting); GRTA9906 60 mg IR capsule (fed)

SUMMARY:
The aim of this clinical study in healthy women is to explore the intestinal uptake (bioavailability) of two different tablets of GRTA9906 (formulations) into the body and the effect of food on it. The intake of food may considerably influence the bioavailability, either by interaction with the compound itself or, if a prolonged release (PR) formulation is used, with the components of the tablet-matrix. For these reasons, the relative bioavailability and the effect of food on the bioavailability of GRTA9906 given as PR tablets compared to immediate release (IR) capsules will be assessed in this study.

During the 4 periods of the study, each participant will receive two 60 mg GRTA9906 PR matrix tablets and two 60 mg GRTA9906 IR capsules under fed conditions (after consumption of a high-fat and high-calorie test meal) and fasting conditions (10 hours before dosing until 4.5 hours after dosing). In each period, the participant will receive the investigational product once.

ELIGIBILITY:
Inclusion Criteria:

* Female Caucasian volunteers aged 18 - 55 years.
* Body mass index between 18 and 29 kilograms per square meter inclusive.
* Good physical and mental health status (no current acute illness) determined on the basis of the medical history and a general clinical examination.
* Normal supine blood pressure (systolic blood pressure greater than or equal to 90 Millimeter mercury (mmHg) and less than or equal to 145 mmHg, diastolic blood pressure greater than or equal to 45mmHg and less than or equal to 90 mmHg) and pulse (greater than or equal to 45 and less than or equal to 90 beats per minute).
* Electrocardiogram (12 lead) considered as normal by the Investigator.
* Results of laboratory tests within the normal ranges for the testing laboratory. The Investigator may include a participant having values outside the accepted range if, in his/her opinion, these values are of no clinical relevance. The decision will be justified.
* Participants giving written consent to participate in this trial.
* Negative pregnancy test (females of childbearing potential only).
* Adequate contraception (females of childbearing potential only; adequate contraception is defined as any form of hormonal contraception or intra-uterine device that needs to be in place for a period of at least 2 months prior to screening. Additional barrier contraception must be used for the duration of the study, defined as from the time of screening to the post-study medical examination, and for at least one full month thereafter. A single barrier method alone or abstinence alone is not acceptable. Women of non-childbearing potential may be included if surgically sterile or post-menopausal for at least 2 years).
* Must be able to tolerate high-fat and high-calorie study-meal.

Exclusion Criteria:

* Diseases and functional disorders of the gastrointestinal tract, hepatobiliary system, renal system or cardiovascular system including marked repolarisation abnormality (e.g. suspicious or definite congenital long QT syndrome) or co-medication that is known to influence cardiac repolarisation substantially.
* Malignancy.
* History of orthostatic hypotension.
* Positive human immunodeficiency virus HIV1/2-antibodies, hepatitis B surface-antigen (HBs), hepatitis B core-antibodies (HBc), Hepatitis C virus (HCV) antibody tests at the prestudy medical examination.
* Drug allergy.
* Bronchial asthma.
* Participation in another clinical study in the last three months before starting this study (exception: characterisation of metaboliser status).
* Blood donation (more than 100 milliliter) in the last three months before the start of the study.
* Evidence of alcohol, medication or drug abuse.
* Positive drug abuse screening test.
* Extremely unbalanced diet (in the opinion of the investigator).
* Excessive consumption of food or beverages containing caffeine or other xanthines (more than five cups of coffee or equivalent per day).
* Smoking of more than 20 cigarettes per day.
* Known or suspected of not being able to comply with the study protocol.
* Neurotic personality, psychiatric illness, or suicide risk.
* History of seizures or at risk (i.e. head trauma, epilepsy in family anamnesis, unclear loss of consciousness).
* Pregnant or breastfeeding.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2003-10-22 (Actual); Primary Completion 2003-12-11 (Actual); Study Completion 2003-12-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter - AUC0-tz | pre-dose, 5, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 13, 16, 20, and 23 hours post-dose
  Area under the concentration vs. time curve from dosing time to the last measured concentration above the lower limit of quantitation. The concentration of GRTA9906 was determined in the serum samples using a validated HPLC-method with fluorometric detection.
Pharmacokinetic parameter - AUC0-inf | pre-dose, 5, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 13, 16, 20, and 23 hours post-dose
  Total area under the concentration vs. time curve (from dosing time to infinity). The concentration of GRTA9906 was determined in the serum samples using a validated HPLC-method with fluorometric detection.
Pharmacokinetic parameter - tmax | pre-dose, 5, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 13, 16, 20, and 23 hours post-dose
  Time to reach maximum serum concentration. The concentration of GRTA9906 was determined in the serum samples using a validated HPLC-method with fluorometric detection.
Pharmacokinetic parameter - Cmax | pre-dose, 5, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 13, 16, 20, and 23 hours post-dose
  Maximum serum concentration. The concentration of GRTA9906 was determined in the serum samples using a validated HPLC-method with fluorometric detection.
Pharmacokinetic parameter - lag-time (tlag) | pre-dose, 5, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 13, 16, 20, and 23 hours post-dose
  Period of time from the administration of the investigational product to the first measured concentration. The concentration of GRTA9906 was determined in the serum samples using a validated HPLC-method with fluorometric detection.
Pharmacokinetic parameter - t(½,z) | pre-dose, 5, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 13, 16, 20, and 23 hours post-dose
  Apparent terminal half-life. The concentration of GRTA9906 was determined in the serum samples using a validated HPLC-method with fluorometric detection.
Pharmacokinetic parameter - MRT | pre-dose, 5, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 13, 16, 20, and 23 hours post-dose
  Mean residence time. The concentration of GRTA9906 was determined in the serum samples using a validated HPLC-method with fluorometric detection.
Pharmacokinetic parameter - HVD | pre-dose, 5, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 13, 16, 20, and 23 hours post-dose
  Half-value duration. The concentration of GRTA9906 was determined in the serum samples using a validated HPLC-method with fluorometric detection.
Pharmacokinetic parameter - CL/f | pre-dose, 5, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 13, 16, 20, and 23 hours post-dose
  Total clearance. The concentration of GRTA9906 was determined in the serum samples using a validated HPLC-method with fluorometric detection.
Pharmacokinetic parameter - Vz/f | pre-dose, 5, 10, 20, 30, 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 13, 16, 20, and 23 hours post-dose
  Apparent volume of distribution during the terminal phase. The concentration of GRTA9906 was determined in the serum samples using a validated HPLC-method with fluorometric detection.

SECONDARY OUTCOMES:
Pupillometry parameter - Initial diameter (mm) | pre-dose and 1, 2, 3, 4, 5, 6, 7, 8, 10 and 23 hours post-dose
  Diameter in millimeter (mm) before presentation of the light stimulus. Pupillometry will be carried out using a Compact Integrated Pupillograph (CIP) in a darkened room.
Pupillometry parameter - Latency time (sec) | pre-dose and 1, 2, 3, 4, 5, 6, 7, 8, 10 and 23 hours post-dose
  Time in seconds (sec) between begin of the light stimulus and onset of pupil reaction.
Pupillometry parameter - Amplitude (mm) | pre-dose and 1, 2, 3, 4, 5, 6, 7, 8, 10 and 23 hours post-dose
  Difference in millimeter (mm) between initial value and minimum diameter.
Pupillometry parameter - Constriction time (sec) | pre-dose and 1, 2, 3, 4, 5, 6, 7, 8, 10 and 23 hours post-dose
  Time in seconds (sec) between onset of reaction and minimum diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Dept. of Human Pharmacology, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No